CLINICAL TRIAL: NCT02907645
Title: Influenza Vaccine Randomized Educational Trial: Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, Associate Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAR0289
Record Dates: First submitted 2016-09-08; First posted 2016-09-20 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Vaccination; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Local educational (Experimental): Adult patients in this arm receive educational information regarding influenza vaccination based on local data
  Interventions: Behavioral: Local educational information
- National educational (Experimental): Adult patients in this arm receive educational information regarding influenza vaccination based on national data
  Interventions: Behavioral: National educational information
- Usual care (No Intervention): No educational information other than provided as usual care by health care providers

INTERVENTIONS:
Behavioral: Local educational information — Adult patients in this arm receive educational information regarding influenza vaccination based on local data
  Arms: Local educational
Behavioral: National educational information — Adult patients in this arm receive educational information regarding influenza vaccination based on national data
  Arms: National educational

SUMMARY:
Influenza vaccine is recommended as routine care for all individuals who are at least 6 months of age and older. Recently, questions about vaccine safety and concerns for side effects have increased, contributing to both influenza vaccine hesitancy and refusal. In an effort to educate patients, public health entities and physicians give informational handouts in various forms.

However, recent publications have found that pro-vaccine messages can have paradoxical effects on vaccine intentions, therefore further studies on vaccine related public health communication is needed. The purpose of this study is to compare the effectiveness of pro-vaccine messages of local data, pro-vaccine messages of national data, and no educational message on patient's receipt of the influenza vaccine. These results will help to understand the relationship between patient education and the intent to vaccinate and receipt of the influenza vaccine as well as to optimize educational information given to patients regarding the influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* visit to study site at time of intervention

Exclusion Criteria:

* prior receipt of influenza vaccine that season

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who receive influenza vaccination on day of intervention | Day 0
  Receipt of influenza vaccination on the day of the educational intervention

SECONDARY OUTCOMES:
Number of participants who receive Influenza vaccination by the end of the influenza vaccine season | Up to 7 months
  Receipt of influenza vaccination by April 2017

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No